CLINICAL TRIAL: NCT05933785
Title: The Value of Transanal Endoscopic Intersphincteric Resection (taE-ISR) in Extreme Anal Preservation in Ultra-low Rectal Cancer
Brief Title: the Value of Transanal Endoscopic ISR
Status: Completed | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: taE-ISR
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transanal endoscopic ISR
  Interventions: Procedure: transanal endoscopic ISR
- traditional ISR

INTERVENTIONS:
Procedure: transanal endoscopic ISR — perform ISR using laparoscopy through transanal port
  Groups: transanal endoscopic ISR

SUMMARY:
The Intersphincteric resection (ISR) technique is an alternative for anal preservation in ultra-low rectal cancer. The transanal total mesorectal excision (TaTME) technique might compensate for the deficiencies of ISR in terms of tumor spillage and poor surgical field exposure. Thus, the investigators perform ISR through a transanal endoscopic approach (taE-ISR), seeking to evaluate the value of this innovative technique in anal preservation in ultra-low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* American Society of Anesthesiologists (ASA) score I to III
* A biopsy proven histological diagnosis of rectal carcinoma
* preoperative stage as (y) cT1-3N0-2M0
* lower margin of the tumor less than 5cm from the anus
* tumor diameter ≤5cm

Exclusion Criteria:

* Pregnant or lactating women
* Synchronous rectal carcinoma
* History of colorectal cancer or other malignant tumors
* Clinical evidence of metastasis
* Emergency procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with low and ultra-low rectal cancer
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
anal preservation rate | 1 year after sugery
  No conversion to APR and closure was closed within 1 year after surgery

SECONDARY OUTCOMES:
incidence of Defecation disorders | 6 months after surgery
  A Wexner score >10 indicated the existence of defecation dysfunction
incidence of positive distal resection margin | 30 days after surgery
  A positive distal resection margin (DRM) was diagnosed with the presence of tumor cells within 1mm from the DRM

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai
  - Shanghai Minimally Invasive Surgery Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided